CLINICAL TRIAL: NCT01600534
Title: GooDMomS: A Multimodel Pregnancy and Postpartum Intervention for Gestational Diabetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-0810
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Gestational Diabetes Mellitus; Pregnancy
Keywords: gestational diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Experimental): Participants obtain access to an internet-based educational intervention.
  Interventions: Behavioral: lifestyle counseling
- Usual Care Lifestyle counseling (Other): Self directed educational intervention
  Interventions: Behavioral: lifestyle counseling

INTERVENTIONS:
Behavioral: lifestyle counseling — Participants receive lifestyle counseling on healthy eating and physical activity through an internet-based program or self-directed educational program.
  Other Names: healthy lifestyle; glucose control

SUMMARY:
This study includes a behavioral educational intervention that focuses on healthy eating and physical activity during pregnancy and the postpartum among women newly diagnosed with gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
This is a pilot trial in which 30 women newly diagnosed with gestational diabetes are randomized to either one of two groups: 1) active internet intervention or 2) self-directed educational intervention. The primary pregnancy outcome is change in A1C. The primary postpartum outcome is weight.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gestational diabetes
* Planning to delivery with the study area

Exclusion Criteria:

* Pre-existing diabetes (type 1 or type 2 diabetes)
* Non-English speaking
* Not planning to delivery in the study area

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin | Baseline and 36 weeks gestation

SECONDARY OUTCOMES:
Change in weight after pregnancy | 6 weeks postpartum to 24 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Nicholson, MD MPH MBA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina clinics, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Setse R, Grogan R, Cooper LA, Strobino D, Powe NR, Nicholson W. Weight loss programs for urban-based, postpartum African-American women: perceived barriers and preferred components. Matern Child Health J. 2008 Jan;12(1):119-27. doi: 10.1007/s10995-007-0211-6. Epub 2007 Jun 7. PMID 17554614
- [Derived] Nicholson WK, Beckham AJ, Hatley K, Diamond M, Johnson LS, Green SL, Tate D. The Gestational Diabetes Management System (GooDMomS): development, feasibility and lessons learned from a patient-informed, web-based pregnancy and postpartum lifestyle intervention. BMC Pregnancy Childbirth. 2016 Sep 21;16(1):277. doi: 10.1186/s12884-016-1064-z. PMID 27654119